CLINICAL TRIAL: NCT04002752
Title: A Double-blind, Placebo-controlled, Randomized, Parallel, Single Dose Study to Investigate Pharmacokinetics, Safety, and Tolerability of JNJ-73763989 in Healthy Japanese Adult Participants
Brief Title: A Study of JNJ-73763989 in Healthy Japanese Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Sciences Ireland UC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CR108646; 2019-000629-31 (EudraCT Number); 73763989HPB1001 (Other: Janssen Sciences Ireland UC)
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Panel A: JNJ-73763989 or Placebo (Experimental): Participants will receive JNJ-73763989 (Dose Level 1) or matching placebo as single subcutaneous injection.
  Interventions: Drug: JNJ-73763989; Drug: Placebo
- Panel B: JNJ-73763989 or Placebo (Experimental): Participants will receive JNJ-73763989 (Dose Level 2) or matching placebo as single subcutaneous injection.
  Interventions: Drug: JNJ-73763989; Drug: Placebo
- Panel C: JNJ-73763989 or Placebo (Experimental): Participants will receive JNJ-73763989 (Dose Level 3) or matching placebo as single subcutaneous injection.
  Interventions: Drug: JNJ-73763989; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-73763989 — Participants will receive JNJ-73763989 as single subcutaneous injection.
Drug: Placebo — Participants will receive placebo matching to JNJ-73763989 as single subcutaneous injection.

SUMMARY:
The purpose of this study is to investigate the pharmacokinetics, safety, and tolerability of JNJ-73763989 in healthy Japanese adult participants following single-dose subcutaneous administration of 3 different doses of JNJ-73763989, Dose Level 1 (Panel A), Dose Level 2 (Panel B) or Dose Level 3 (Panel C).

ELIGIBILITY:
Inclusion Criteria:

* Participant must be a Japanese participant who has resided outside Japan for no more than 10 years and whose parents and grandparents are Japanese, as determined by participant's verbal report
* Participant must have a body mass index (BMI; weight in kilogram [kg] divided by the square of height in meters) of 18.0 to 30.0 kilogram per square meter (kg/m^2) extremes included, and body weight not less than 45.0 kg
* Participant must be healthy on the basis of physical examination, clinical laboratory tests, medical history, and vital signs performed at screening. In case of abnormalities (except for those listed in the exclusion criteria) a participant may be included after all if the investigator judges the abnormalities not clinically significant or appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* A female participant of childbearing potential must have a negative highly sensitive serum (beta-human chorionic gonadotropin [beta-hCG]) at screening and a negative urine pregnancy test on Day -1
* A male participant must agree not to donate sperm after enrollment (Day 1) in the study until at least 90 days after receiving the study drug

Exclusion Criteria:

* Participant with a history of cardiac arrhythmias (for example, premature ventricular contractions), history of risk factors for Torsade de Pointes syndrome (for example, hypokalemia, family history of long QT Syndrome)
* Female participant who is pregnant, breast-feeding, or planning to become pregnant during the study or within 90 days after receiving the study drug (or longer, if dictated by local regulation)
* Male participants who plan to father a child during the study or within 90 days after receiving the study drug (or longer, if dictated by local regulation)
* Participant with human immunodeficiency virus type 1 (HIV-1) or type 2 (HIV-2) infection (confirmed by antibodies) at screening
* Participant with current hepatitis A infection (confirmed by hepatitis A antibody immunoglobulin M [IgM]), or hepatitis B infection (confirmed by Hepatitis B surface antigen [HBsAg]), or hepatitis C virus (HCV) infection (confirmed by HCV antibody), or hepatitis E infection (confirmed by hepatitis E antibody IgM) at screening

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2019-08-23 (Actual); Study Completion 2019-08-23 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of JNJ-73763989 | Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, and 48 hours postdose
  Cmax is the maximum observed plasma analyte concentration.
Time to Reach Maximum Observed Plasma Concentration (Tmax) of JNJ-73763989 | Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, and 48 hours postdose
  Tmax is defined as actual sampling time to reach maximum observed plasma analyte concentration.
Last Measurable Observed Plasma Concentration (Clast) of JNJ-73763989 | Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, and 48 hours postdose
  Clast is last measurable observed plasma analyte concentration.
Area Under the Plasma Concentration-Time Curve from Time Zero to the Time of the Last Measurable Concentration (AUC[0-last]) of JNJ-73763989 | Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, and 48 hours postdose
  AUC(0-last) is area under the plasma concentration-time curve from time zero to the time of the last measurable (non-below quantification limit [non-BQL]) concentration, calculated by linear-linear trapezoidal summation.
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to 30 days after last study drug administration (Up to 7 weeks)
  AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Sciences Ireland UC Clinical Trial, Study Director — Janssen Sciences Ireland UC
Locations (1):
- PAREXEL International, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Gane E, Yuen MF, Kakuda TN, Ogawa T, Takahashi Y, Goeyvaerts N, Lonjon-Domanec I, Vaughan T, Schluep T, Hamilton J, Njumbe Ediage E, Hillewaert V, Snoeys J, Lenz O, Talloen W, Biermer M. JNJ-73763989 pharmacokinetics and safety: Liver-targeted siRNAs against hepatitis B virus, in Japanese and non-Japanese healthy adults, and combined with JNJ-56136379 and a nucleos(t)ide analogue in patients with chronic hepatitis B. Antivir Ther. 2022 Jun;27(3):13596535221093856. doi: 10.1177/13596535221093856. PMID 35695169